CLINICAL TRIAL: NCT00327834
Title: Atomoxetine in the Treatment of Binge Eating Disorder: A Single-Center, Double-Blind, Placebo-Controlled, Flexible Dose Study in Outpatients
Brief Title: Atomoxetine in the Treatment of Binge Eating Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Susan McElroy, Lindner Center of HOPE
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B4Z-US-X009
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Binge-eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine

SUMMARY:
The specific aim of this study is to assess the efficacy and safety of atomoxetine compared with placebo in outpatients with binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet the DSM-IV criteria for a diagnosis of binge-eating disorder for at least the last 6 months
* In addition, subjects will report at least 3 binge eating episodes per week for the last 6 months prior to randomization

Exclusion Criteria:

* Have concurrent symptoms of bulimia nervosa or anorexia nervosa
* Women who are pregnant, lactating, or of child bearing potential who are not using adequate contraceptive measures
* Patients who are displaying clinically significant suicidality or homicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L: McElroy, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Guerdjikova A, Kotwal R, Welge JA, Nelson EB, Lake KA, Keck PE Jr, Hudson JI. Atomoxetine in the treatment of binge-eating disorder: a randomized placebo-controlled trial. J Clin Psychiatry. 2007 Mar;68(3):390-8. doi: 10.4088/jcp.v68n0306. PMID 17388708